CLINICAL TRIAL: NCT04232150
Title: Midazolam's Anterograde Amnesia Efficacy in Noisy Orthopedic Surgery: Does Midazolam Cause Effective Anterograde Amnesia in Noisy Orthopedic Surgeries?
Brief Title: Does Midazolam Cause Effective Anterograde Amnesia in Orthopedic Surgeries?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Abdelkarim S. Aloweidi (Unknown)
Responsible Party: Principal Investigator, Mahmoud M. Almustafa, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 67/2019/865
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia; Orthopedic Surgery
Keywords: Midazolam; Orthopedic surgery; total knee replacement; total hip replacement
MeSH Terms: interventions — Midazolam; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Overall, 116 patients were enrolled, out of which 20 were excluded before start of study for the following reasons: contraindication for spinal anesthesia (n=10), preoperative administration of sedative agent (n=3), refusal to be enrolled in study (n=4), a patient with neurological disorder (Schizophrenia), a blind patient, and a deaf patient. Of the 96 patients included, 33 were enrolled in group C, 32 in group S; however, 2 patients requested a deeper level of sedation so an added dose of midazolam and fentanyl were given thus excluding them from study, and 31 patients in group R.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (control group) (Experimental): control group will receive no sedation under spinal anesthesia.
  Interventions: Procedure: spinal anesthesia with no sedation.
- Group O (single dose group) (Experimental): patients will receive 0.025mg/kg midazolam sedation under spinal anesthesia.
  Interventions: Drug: single-dose midazolam for sedation under spinal anesthesia.
- Group M (double dose group) (Experimental): patients will receive 0.025mg/kg midazolam sedation twice under spinal anesthesia.
  Interventions: Drug: Double-dose midazolam for sedation under spinal anesthesia.

INTERVENTIONS:
Drug: single-dose midazolam for sedation under spinal anesthesia. — Induction of neuraxial anesthesia was done using 2.8cc of 0.5 % Heavy Bupivacaine and 20mcg fentanyl injected intrathecally for all patients. Supplemental oxygen was given via facemask with capnography monitoring. Group O received 0.025mg/kg midazolam at skin incision.
  Arms: Group O (single dose group)
Drug: Double-dose midazolam for sedation under spinal anesthesia. — Induction of neuraxial anesthesia was done using 2.8cc of 0.5 % Heavy Bupivacaine and 20mcg fentanyl injected intrathecally for all patients. Supplemental oxygen was given via facemask with capnography monitoring. Group M received 0.025mg/kg midazolam at skin incision and repeated 5 minutes before maximum stimulation.
  Arms: Group M (double dose group)
Procedure: spinal anesthesia with no sedation. — Induction of neuraxial anesthesia was done using 2.8cc of 0.5 % Heavy Bupivacaine and 20mcg fentanyl injected intrathecally for all patients. Supplemental oxygen was given via facemask with capnography monitoring.
  Arms: Group C (control group)

SUMMARY:
Spinal anesthesia is one of the commonest choices of anesthesia for infraumbilical surgeries.The use of sedation has markedly increased patients' comfort and acceptance towards spinal anesthesia. The aim of this study is to investigate visual, recall, auditory recall, and sedation scores among patients receiving Midazolam for sedation during spinal anesthesia in patients undergoing orthopedic surgeries.

DETAILED DESCRIPTION:
Spinal anesthesia is one of the commonest choices of anesthesia for infraumbilical surgeries.The use of sedation has markedly increased patients' comfort and acceptance towards spinal anesthesia. The main goals of sedation for surgeries under spinal anesthesia are patient comfort, preservation of protective airway reflexes, and the help in the maintenance of hemodynamic stability during the surgical procedure. The aim of this study is to investigate visual, recall, auditory recall, and sedation scores among patients receiving Midazolam for sedation during spinal anesthesia in patients undergoing orthopedic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee or total hip replacement.
* ASA I, II, or III.
* patients undergoing spinal anesthesia.

Exclusion Criteria:

* patient refusal.
* <24 hours sedative administration.
* patient with hearing impairment.
* neurological or memory disorder.
* abnormal kidney function tests.
* any contraindication for spinal anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative recall of auditory stimuli and intraoperative noise | 4 months
  For auditory recall, a question was asked by the surgeon to the patient at maximum stimulation. Patients were examined for auditory recall by following-up the patients postoperatively in the inpatient department.
Postoperative recall of visual stimuli | 4 months
  For visual recall, a picture of a horse assigned at maximum stimulation, a cat at recovery room, and a bird after discharge to the inpatient department. Patients were examined for visual recall by following-up the patients postoperatively in the inpatient department.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No